CLINICAL TRIAL: NCT05407896
Title: End-Stage Kidney Disease Interactive Decision Aid for the Elderly (myKIDNEY)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Singapore General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Semra Ozdemir, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-SMF-0007
Record Dates: First submitted 2021-07-05; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: End-Stage Kidney Disease
Keywords: end-stage kidney disease; decision aid; shared decision making
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Pre-post study design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison arm (No Intervention): Patients and caregivers in this arm will receive existing counselling by trained counsellors.
- Intervention arm (Experimental): Patients and caregivers in this arm will receive counselling with the newly developed web-based decision aid (myKIDNEY) by trained counsellors.
  Interventions: Other: myKIDNEY decision aid

INTERVENTIONS:
Other: myKIDNEY decision aid — Patients and caregivers will be counselled using myKIDNEY decision aid which includes a video. Patients will be asked to complete a values clarification exercise (VCE). If a caregiver is recruited without their patient, he/she will be asked to complete the VCE on patient's behalf (i.e., surrogate). At the end of VCE, the participant will be given real-time feedback on which treatment might be the best fit for the patient. With the patient's consent, this information will be shared with the treating physician who can then make recommendations based on the patient's preferences.
  Arms: Intervention arm

SUMMARY:
Decision aids are highly recommended for decisions when there is no "right" treatment choice. The goal is to help patients choose a treatment that is consistent with their preferences and to minimize decisional conflict and regret. A case where there is no "right" treatment concerns the decision to undergo dialysis or supportive care (i.e., conservative management) for elderly (aged ≥70) patients with end-stage kidney disease. The investigators propose to develop an interactive web-based decision aid and test its effectiveness via a pre-post study design. This research aims to reduce decisional conflict for elderly ESKD patients and caregivers.

DETAILED DESCRIPTION:
For patients aged 75 and above with comorbidities, the benefits of dialysis over kidney supportive care, which focuses on maintaining quality of life as opposed to life extension, are not clear. As there is no clear or "right" treatment choice, treatment decisions should be informed by patient preferences. However, currently in Singapore most patients choose dialysis and express decisional conflict and regret. Decision aids (DAs) together with values clarification methods (VCMs) can help patients choose a treatment that is concordant with their preferences and treatment goals. To help minimize decisional conflict among elderly ESKD patients, the first aim of this proposal is to adapt the current materials the investigators have developed (booklet and video) for elderly ESKD patients in a prior effort (NMRC/HSRG/0080/2017) into an interactive web-based tool called myKIDNEY. It will provide patients with tailored and relevant information based on their age and medical history, and help them identify and express their preferences via an interactive VCM. The second aim of the proposal is to test the benefits of counselling with myKIDNEY to standard renal counselling via a pre-post study design. The primary hypothesis is that patients and caregivers who receive counselling with myKIDNEY will report less decisional conflict compared to those who receive standard counselling. The investigators also hypothesize that fewer patients in the intervention arm will opt for dialysis, which is the more costly and invasive treatment option. If the proposed study shows evidence that the interactive tool improves decision-making quality in the local setting, this will result in a better patient experience. If fewer patients choose dialysis as per our hypothesis, this will also generate cost savings for the health system while at the same time allowing patients to choose their preferred treatment with lower chances of decisional conflict.

ELIGIBILITY:
Inclusion Criteria (patients):

* Incident CKD Stage 5 patients with GFR<15ml/min
* Aged 70 years or older-
* Have not undergone counselling with a renal counsellor
* Cognitively intact as determined by the Abbreviated Mental Test (AMT)
* Speak and read English or Mandarin

Inclusion Criteria (caregivers):

* Primary informal caregiver for an eligible patient (primarily involved in providing care, ensuring provision of care, and/or in making decisions regarding patient's care)
* Aged 21 years and older
* Direct relative of the patient

Exclusion Criteria:

- Patients deemed to be mentally incompetent, and those not aware of their diagnosis will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict scale (0 to 100; higher scores indicate higher decisional conflict) | 1 hour
  Difference in decisional conflict scale between the intervention and comparison arms

SECONDARY OUTCOMES:
Stated preferred treatment | Assessed after renal counselling (within 2 weeks after renal counselling)
  Difference in the percentage of participants who choose a form of dialysis as the preferred treatment between the intervention and comparison arms
Actual treatment choice | 6 months after renal counselling
  Difference in the percentage of participants who initiate dialysis based on the medical records at 6 months after the counselling between the intervention and comparison arms
Actual treatment choice | 12 months after renal counselling
  Difference in the percentage of participants who initiate dialysis based on the medical records at 12 months after the counselling between the intervention and comparison arms

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request.